CLINICAL TRIAL: NCT05056480
Title: Learning Health for Pediatric Complex Care Integration (PCCI)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00104642
Record Dates: First submitted 2021-09-20; First posted 2021-09-24 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2021-09

CONDITIONS: Children and Youth With Special Healthcare Needs; Care Coordination
Keywords: Care coordination; Complex care; Interdisciplinary care
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents/caregivers: Parents/caregivers of children <20 years old who received interdisciplinary care coordination within the Pediatric Complex Care Integration (PCCI) program
  Interventions: Other: Surveys
- Clinical staff: PCCI care management staff participating in implementation of the PCCI program
  Interventions: Other: Surveys

INTERVENTIONS:
Other: Surveys — Parent/caregivers participants will complete multiple repeating surveys to gather family-reported perspectives on the impact of the PCCI care management program. Clinical staff participants will complete multiple repeating surveys that gather clinician perspectives on the impact of the PCCI care management program. Parent/caregiver and clinical staff participants will also be invited to participated in one-on-one semi-structured interviews with the study team.
  Other Names: Interviews

SUMMARY:
The study team will conduct a mixed methods evaluation of the implementation of an evidence-based clinical program -- the Pediatric Complex Care Integration (PCCI) program - for improvement of care integration for children and youth with special healthcare needs (CYSHCN) and children with medical complexity (CMC). The PCCI program is not a discrete intervention itself; rather it is a health system-initiated program that will be implemented as a new standard of care for eligible patients with the intention of improving quality of care, implemented by clinical teams within Duke Health.

ELIGIBILITY:
* Inclusion criteria for children and parents/caregivers:

  * Patients up to 20 years old or under at the time of the monthly data pull or clinical team recommendation (for participation in the PCCI clinical program; no minors under 18 years old will be directly surveyed)
  * Adult parents/caregivers of participating children (for participation in interviews and quantitative parent-reported surveys) *For human-centered design interviews, PCCI program participation is not required
  * Primary care attributed to Duke Pediatrics Primary Care - Roxboro Road clinic
  * High level of medical complexity: CSHCN (level 2 PMCA) or CMC (level 3 PMCA)
  * High risk for future healthcare utilization - may be defined by provider/care team determination, EHR data-based risk prediction model (exempt IRB Pro00104983, Developing a Model to Predict Risk for Healthcare Utilization by Children with Chronic Conditions), or any other way in which the clinical team determines a patient is "high risk" as part of their standard practice/care.
* Exclusion criteria for children and parents/caregivers: children/parents will be excluded if they meet the below criteria:

  * Unable to provide informed consent
  * Non-English or Spanish speaking parent/caregiver or young adult patient
* Inclusion criteria for clinical staff and providers (participation in interviews and quantitative staff/provider-reported surveys):

  * Currently employed by Duke Health
  * Primary site of work at participating primary care clinic site or central DUHS PHMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult parents/caregivers of children/youth who have primary care attributed to Duke Pediatrics Primary Care - Roxboro Road clinic and are receiving complex care management within the PCCI clinical program.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in care fragmentation, as measured by the Pediatric Integrated Care Survey (PICS) | Baseline, 6 months, 12 months
  The PICS is a 20-item survey that gathers parents perspectives on the degree of care integration received by their child using a 6-level Likert scale (1=never; 6=always).
Change in child health-related quality of life (HR-QOL), as measured by the PROMIS (7+2) Parent Proxy Global Health Survey | Baseline, 3 months, 6 months, 9 months, 12 months
  The PROMIS (7+2) Pediatric Global Health Survey is a 9-item parent-reported survey that gathers parent perspectives on their child's overall HR-QOL. Four of the 9 survey items use a 5-level Likert scale with 1=poor and 5=excellent; three of the 9 survey items use a 5-level Likert scale with 1=never and 5=always; and three of the 9 survey items use a 5-level Likert scale with 1=never and 5=almost always.
Change in parent health-related quality of life (HR-QOL), as measured by the PROMIS Global Health Survey | Baseline, 3 months, 6 months, 9 months, 12 months
  The PROMIS Global Health Survey is a 10-item parent-reported survey that gathers parent perspectives on their own overall HR-QOL. Six of the 9 survey items use a 5-level Likert scale with 1=poor and 5=excellent; one of the 9 survey items uses a 5-level Likert scale with 1=not at all and 5=completely; one of the 9 survey items uses a 5-level Likert scale with 1=never and 5=always; one of the 9 survey items uses a 5-level Likert scale with 1=none and 5=very severe; and one of the 9 survey items uses a 0-10 scale (0=no pain; 10=worst pain imaginable).
Change in well-being, as measured by the Well-Being Index (WBI) | Baseline, 3 months, 6 months, 12 months
  The Well-Being Index is a 9-time clinical provider/staff-reported measure that gathers staff perceptions of their overall well-being at work. Seven of the 9 survey items use a dichotomous response (Yes/No) and two remaining items use 7-level Likert scale (1=very strongly disagree; 7=very strongly agree).

SECONDARY OUTCOMES:
Change in caregiver self-management, as measured by the Parent-Patient Activation Measure (P-PAM) | Baseline, 3 months, 6 months, 12 months
  The Parent-Patient Activation Measure (P-PAM) is a 13-item parent-reported survey that uses a 4-level Likert scale (1=disagree strongly; 4=agree strongly).
Change in perceptions of barriers to care, as measured by the Barriers to Care Questionnaire (BCQ) | Baseline, 12 months
  The 19-item Barriers to Care Questionnaire (BCQ) gathers parent perspectives on barriers encountered when trying to get health care for their child. The BCQ uses a 5-level Likert scale (0=never; 4=almost always).
Change in perceptions of cultural distance, as measured by the Cultural Distance Scale (CDS) | Baseline, 12 months
  The 4-item Cultural Distance Scale (CDS) is a parent-reported survey that uses a 6-level Likert scale (1=very similar; 6=very different).
Changes in caregiver self-efficacy, as measured by the New Generalized Self-Efficacy Scale (NGSE) | Baseline, 3 months, 6 months, 9 months, 12 months
  The 8-item New Generalized Self-Efficacy Scale is a parent-reported survey uses a 5-level Likert scale (1=strongly disagree; 5=strongly agree).
Changes in perceptions of shared decision-making, as measured by the a sub-scale from the Interpersonal Processes of Care survey | 3 months, 6 months, 9 months, 12 months
  This 4-item sub-scale from the Interpersonal Processes of Care survey focuses on perceptions of shared-decision making. Parents respond to questions on a 5-level Likert scale (1=never; 5=always).
Feasibility, as measured by clinical staff survey | 12 months
  Perceptions of the feasibility of implementation of the PCCI care management program, as measured by the Feasbility of Intervention Measure (FIM)
Acceptability, as measured by clinical staff survey | 12 months
  Perceptions of the acceptability of implementation of the PCCI care management program, as measured by the Acceptability of Intervention Measure (AIM)
Appropriateness, as measured by clinical staff survey | 12 months
  Perceptions of the appropriateness of implementation of the PCCI care management program, as measured by the Intervention Appropriateness Measure (IAM)

CONTACTS AND LOCATIONS:
Overall Officials: David Y Ming, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No